CLINICAL TRIAL: NCT03658759
Title: ECPR Treatment Protocol: Rapid Response VA-ECMO in Refractory Out-of-hospital Cardiac Arrest (RESuSCITATe Registry)
Brief Title: Rapid Response VA-ECMO in Refractory Out-of-hospital Cardiac Arrest
Acronym: RESuSCITATe
Status: Withdrawn | Type: Observational
Why Stopped: Study cancelled
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, J.P.S Henriques, Prof. dr. J.P.S. Henriques, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: ECPR-062018-UAMC
Record Dates: First submitted 2018-06-27; First posted 2018-09-05 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Out-Of-Hospital Cardiac Arrest
Keywords: Extra corporeal Life support; extracorporeal cardiopulmonary resuscitation; refractory out-of-hospital cardiac arrest; extra corporeal membrane oxygenation; mechanical circulatory support; mechanical chest compressions
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest | interventions — Ex utero Intrapartum Treatment Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Extracorporeal Cardiopulmonary Resuscitation — local ECPR clinical pathway, including transport with mechanical chest compression device and rapid response VA-ECMO
  Other Names: Extra Corporeal Life support; Extra Corporeal Membrane Oxygenation; Mechanical chest compressions

SUMMARY:
A selected group of patients with refractory cardiac arrest may benefit from inhospital treatment and this may warrant transfer to the hospital with ongoing CPR. In patients with VF or ventricular tachycardia (VT) the underlying cause may be reversible and damage to other organs is limited at the time of the arrest. Many patients will have a coronary event that can be treated by angioplasty. However, up to now absence of ROSC poses a barrier for angioplasty, and most patients are therefore not even transported to a hospital. With the use of extra corporeal membrane oxygenation (ECMO) the circulation can be restored immediately, providing time to diagnose and treat the underlying cause of the cardiac arrest. International cohort studies show that a strategy of pre-hospital triage and transport to a cardiac arrest expertise center for "rapid-response" ECMO and coronary revascularization is feasible and improves survival.

A clinical pathway will encompass intense cooperation and optimal logistics between several paramedical and medical disciplines, i.e. from prehospital ambulance service to intensive care. Incorporation of mechanical chest compressions devices (LUCAS™), rapid-response veno-arterial (VA-)ECMO (Cardiohelp, Maquet), and ECMO assisted revascularization in a dedicated clinical pathway will offer a potential lifesaving treatment option that is in accordance with the recommendations in the current Guidelines.

The aim of the study is to investigate the feasibility of a new local clinical pathway in our hospital to provide ECPR for refractory OHCA patients.

DETAILED DESCRIPTION:
Coronary heart disease is the leading cause of cardiac arrest. The incidence of cardiac arrest in Europe is between 0.4 and 1 per 1000 inhabitants per year, thus involving between 350.000 and 700.000 people per year. Approximately, 275.000 of these cardiac arrests are treated by the emergency medical service (EMS) in Europe. (1) Survival after cardiac arrest varies from less than 5% to 60% according to the characteristics of the cardiac arrest event (e.g. cardiac etiology, witnessed arrest, initial recorded rhythm (shockable: ventricular fibrillation (VF), ventricular tachycardia (VT) or not shockable).(1) Cardiac arrest patients, who despite conventional cardiopulmonary resuscitation (CPR) do not achieve return of spontaneous circulation (ROSC) within 10-20 minutes of advanced life support (ALS) have the worst prognosis with rates of survival to hospital discharge of 2-11%.

A selected group of patients with refractory cardiac arrest may benefit from very aggressive in-hospital treatment and this may warrant transfer to the hospital with ongoing CPR. In patients with VF or ventricular tachycardia (VT) the underlying cause may be reversible and damage to other organs is limited at the time of the arrest. Many patients will have a coronary event that can be treated by angioplasty. However, up to now absence of ROSC poses a barrier for angioplasty, and most patients are therefore not even transported to a hospital.

With the use of extra corporeal membrane oxygenation (ECMO) the circulation can be restored immediately, providing time to diagnose and treat the underlying cause of the cardiac arrest. International cohort studies show that a strategy of pre-hospital triage and transport to a cardiac arrest expertise center for "rapid-response" ECMO and coronary revascularization is feasible and improves survival. The recent 2015 European Resuscitation Council Guidelines for Resuscitation position extracorporeal CPR (ECPR) as follows: "ECPR should be considered as a rescue therapy for those patients in whom initial advanced life support (ALS) measures are unsuccessful and to facilitate specific interventions (e.g. coronary angiography and percutaneous coronary intervention (PCI) or pulmonary thrombectomy for massive pulmonary embolism)".(2) A recent meta-analysis performed by our group supports ECMO in this setting. (3)

Currently, a strong pre-hospital and clinical pathway for acute myocardial infarction exists in the greater Amsterdam region / Noord-Holland region, i.e. "Lifenet protocol". The Academic Medical Center is an international recognized center with the ARREST program to evaluate treatments for out-of-hospital cardiac arrest (OHCA).(4) However, a dedicated clinical pathway for refractory OHCA patients does not yet exist. Integration of the "Lifenet protocol" and ARREST program would provide an ideal setting to create and install a dedicated clinical pathway for these cardiac arrest patients.

The existing clinical pathway for cardiac arrest patients will be optimized and upgraded to be able to provide ECPR for refractory cardiac arrest patients. This clinical pathway will encompass intense cooperation and optimal logistics between several paramedical and medical disciplines, i.e. from pre-hospital ambulance service to intensive care. Incorporation of mechanical chest compressions devices (LUCAS™), rapid-response veno-arterial (VA-)ECMO (Cardiohelp, Maquet), and ECMO assisted revascularization in a dedicated clinical pathway will offer a potential lifesaving treatment option that is in accordance with the recommendations in the current Guidelines.

The aim of the study is to investigate the feasibility of a new local clinical pathway to provide ECPR for refractory OHCA patients.

ELIGIBILITY:
Inclusion Criteria:

* Witnessed arrest
* Bystander CPR initiated before EMS arrival or EMS-witnessed arrest
* VF/VT as first recorded rhythm by EMS or shock delivered by AED
* No ROSC within 10 minutes after EMS arrival
* Ambulance transport with mechanical chest compression device

Exclusion Criteria:

* Confirmation of ROSC
* End-tidal CO2 < 10 mmHg
* Known terminal disease (eg. cancer)
* Known severe comorbidity

  * Severe chronic pulmonary disease (GOLD classification 3 or 4)
  * Heart failure NYHA classification 3 or 4
  * Known history of bifemoral surgery
* Do Not Resuscitate (DNR) order
* Expected time from transport decision to start ECMO >60 minute

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with refractory OHCA due to VF/VT, witnessed cardiac arrest and basic life support before EMS arrival.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-07-02 (Actual); Primary Completion 2019-12-02 (Estimated); Study Completion 2020-07-02 (Estimated)

PRIMARY OUTCOMES:
1-year mortality | assessed through study completion: at 1-year.

SECONDARY OUTCOMES:
Adverse outcomes | assessed through study completion: for the time in the hospital , at 30-days and at 1-year.
  Major adverse cardiac events (MACE) (death, myocardial infarction, revascularization, stent thrombosis, stroke, bleeding)
  * CPR-related complications (chest wall compartment syndrome, pneumothorax, chylothorax, pulmonary hemorrhage)
  * ECMO-related complications (bleeding requiring transfusion or surgery, stroke, sepsis, limb ischemia requiring intervention, system or cannula change)
  * Other complications (acute renal failure, ulcer bleeding, pneumonia, sepsis)
Other clinical endpoints: Mortality rate - patients not treated with ECPR in comparison to patients treated with ECPR | assessed through study completion: at 30-days, at 1-year after inclusion of patient
  Mortality rate of patients treated with ECPR in comparison to refractory OHCA patients treated outside of the hours in which ECPR can take place
Percentage of successful cannulations | assessed through study completion: at 1 year and at the end of study inclusion period (expected to be at 1.5 years)
Neurological outcome at 6 months on the cerebral performance category scale (CPC) | assessed through study completion: at 6 months after inclusion of patient.
  measured with CPC scale: CPC 1A return to normal cerebral function and normal living CPC 2 Cerebral disability but sufficient function for independent activities of daily living CPC 3 Severe disability, limited cognition, inability to carry out independent existence CPC 4 Coma CPC 5 Brain death
Quality of life at 6 months assessed by Short form 36 (SF-36) | assessed through study completion: at 6 months after inclusion of patient.
  measured with quality of life assesment form Short form 36 (SF-36). The SF-36 comprises 36 items and contains eight subscales: physical functioning, social functioning, physical role functioning, emotional role functioning, mental health, vitality, bodily pain and general health. Scores are expressed on a scale of 0-100, higher values indicate better quality of life and wellbeing.
Rate of eligible / ineligible patients treated with ECPR | assessed through study completion: at 1 year and at the end of study inclusion period (expected to be at 1.5 years)
  How many patients that were treated with ECPR were retrospectively eligible for treatment with ECPR, in comparison to how many patients were treated, but not eligible.
Noted reasons for non-adherence to the eligibility criteria ECPR | assessed through study completion: at 1 year and at the end of study inclusion period (expected to be at 1.5 years)
  If patients were treated with ECPR, but were not eligible, what were reasons to do so? (for instance: no knowledge beforehand of ineligibility, or, knowledge beforehand of ineligibility but expert decision to treat, etc.)
Number of patients with complete data collection | assessed through study completion: at 1 year and at the end of study inclusion period (expected to be at 1.5 years)
Rate of eligible / ineligible patients not treated with ECPR | assessed through study completion: at 1 year and at the end of study inclusion period (expected to be at 1.5 years)
  How many patients that were not treated with ECPR were retrospectively eligible for treatment with ECPR, in comparison to how many patients were not treated, and not eligible.
30-days mortality | assessed through study completion: at 30-days

CONTACTS AND LOCATIONS:
Overall Officials: Jose P.S. Henriques, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Academic Medical Center, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided